CLINICAL TRIAL: NCT05965661
Title: A New 3D Virtual Reality-based Upper Limb Training to Improve Dexterity in Parkinson's Disease: a Randomized Pilot Study
Brief Title: A New 3D Virtual Reality-based Upper Limb Training to Improve Dexterity in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-01545
Record Dates: First submitted 2023-07-13; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; virtual reality training; dexterity; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: Randomized pilot study
Who Masked: Outcomes Assessor
Masking Description: VR upper limb hand training or VR control training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality upper limb hand training (Other): The PD patients randomized in the experimental group will receive virtual reality upper limb hand training.
  Interventions: Other: virtual reality upper limb hand training
- Virtual reality control training (Other): The PD patients randomized in the control group will receive virtual reality control training.
  Interventions: Other: virtual reality control training

INTERVENTIONS:
Other: virtual reality upper limb hand training — The PD patients randomized in the experimental group will receive virtual reality upper limb hand training.
  Arms: Virtual reality upper limb hand training
Other: virtual reality control training — The PD patients randomized in the control group will receive virtual reality control training.
  Arms: Virtual reality control training

SUMMARY:
We investigate the impact of a 4-week virtual reality-based upper limb training in Parkinson's disease. The benefits on dexterity of this training program will be evaluated.

For these purposes, a randomised, two arm, single assessor blind, parallel design with a monocentric, study setup will be performed.

DETAILED DESCRIPTION:
Patients with Parkinson's disease (PD) suffer from significantly decreased coordination and have difficulties with precise hand/finger movements during the performance of both basic activities of daily living (ADL), such as dressing, grooming as well as higher ADL, such as cooking, shopping and regular medication intake. These difficulties further add to the burden of the disease, leading to reduced quality of life (QoL). A relatively new, but rapidly growing aspect of training in PD neurorehabilitation offers virtual reality (VR). We explore the effects of a VR-based upper limb hand training compared to a VR control training, which is less specific for dexterity. Moreover, we examine the effetcs of the trainings on upper limb related ADL, and therefore the impact on QoL in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed PD, according to UK Brain bank Criteria
* Hoehn & Yahr Stadium I to IV
* Age 40 to 99 years
* written and signed informed consent
* self-reported dexterous difficulties

Exclusion Criteria:

* MoCA <21/30
* psychiatric disease
* participation on other interventional trials
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* severe visual impairment

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
fine finger movements | 4 weeks
  Coin rotation task (CRT): The CRT measures fine coordinated finger movements and is a suitable and valid dexterity test in patients with PD. The seconds for 20 halfturns will be measured.

SECONDARY OUTCOMES:
hand dexterity | 4 weeks
  Nine Hole Peg test (9-HPT): The 9-HPT is a standardized, well established, and reliable measure of hand dexterity in patients with PD. seconds will be measured.
grip strenght | 4 weeks
  The handheld JAMAR dynamometer measures the grip strength. kg will be measured.
motor function | 4 weeks
  MDS-Sponsored Revision of the Unified Parkinson Disease Rating Scale (MDS-UPDRS III): It evaluates motor aspects of Parkinson's disease
self-reported dexterity related problems in daily living | 4 weeks
  Dexterity Questionnaire 24 (DextQ-24): This questionnaire is a standardized patient self-rated outcome measure (PROM) for evaluating dexterity related ADL in PD. score range 24-96, higher scores mean more dexterity problems.
self-reported problems in quality of life | 4 weeks
  Parkinson's Disease Questionnaire (PDQ-39): This questionnaire is a standardized patient self-rated outcome measure (PROM) for evaluating QOL in PD. range 0-156, higher values mean more problems.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanbellingen, Prof, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No